CLINICAL TRIAL: NCT04928443
Title: The Management of Surgical Scars Around Knee After Pediatric Orthopedic Surgery: an Observational, Case-control Study.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202100112B0A3
Record Dates: First submitted 2021-06-14; First posted 2021-06-16 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-06

CONDITIONS: Surgical Scar
Keywords: Scar-care; Surgical wound; Incision site; Cicatrix; Fibrosis; Knee; Pediatric; Orthopedic Procedures
MeSH Terms: conditions — Surgical Wound; Cicatrix; Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Scar dressing group: Patients planning to treat surgical scar with scar dressing
  Interventions: Other: Scar dressing group
- Regular care group: Patients treated with adhesive tapes or strips or did not take care of surgical scar.
  Interventions: Other: Regular care group

INTERVENTIONS:
Other: Scar dressing group — Patients treated with scar dressing for surgical scar care are invited to participate this study and allocated in scar dressing group despite the length of caring period.
  Groups: Scar dressing group
Other: Regular care group — Patients receiving regular scar care are retrospectively identified with matching factors, such as gender, age, length of surgical wound and surgical procedure.
  Groups: Regular care group

SUMMARY:
Scar is an unpleasant symptom that commonly appear after orthopedic surgery, especially the joint procedure. Due to the wide motion range, skin around joint has excessive tension that may increase risk for wide or conspicuous scar formation of surgical wound. Noticeable scar can negatively impact the quality of life and psychosocial development. However, scar management is overlooked in early recovery period easily. Patients commonly start to turn their attention to the surgical scar after the completion of rehabilitation or the resolution of disease or unbearable symptom. It is always beyond the best period of scar treatment, 3 to 6 months after wound healing. This study is aimed to observe and evaluate the scar formation with or without aggressive management in pediatric population within 6 months after wound healing.

DETAILED DESCRIPTION:
This is an observational, case-control study. Patients will be invited to participate and allocated to scar dressing group if they plan to use scar dressing. After gaining the written inform consent, participants will be asked to fulfill the patient diary, including the record of scar dressing use, patient scar assessment scale and satisfaction assessment, with parents' help. In regular group, patients are retrospectively selected by matched factors, such as demographics data. Scar-related data, including scar pictures, vancouver scar scale assessment and complication, are collected from medical history in both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 5 to 18 years
2. Had orthopedic surgery 3 weeks ago and within 6 weeks
3. Had incision sites around the knee
4. All surgical wounds healed completely
5. Length of surgical wounds between 2 and 15 centimeters
6. Planed to treat incisional scar with scar dressing, adhesive tapes, or adhesive strips

Exclusion Criteria:

1. Surgical wound infection
2. Atopic dermatitis or sensitive skin
3. Not able to make return visits regularly
4. Participation was not appropriate determined by physician

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 1. Patients aged 5 to 18 years
  2. Had orthopedic surgery 3 weeks ago and within 6 weeks
  3. Had incision sites around the knee
  4. All surgical wounds healed completely
  5. Length of surgical wounds between 2 and 15 centimeters
  6. Planning to treat incisional scar with scar dressing, adhesive tapes, or adhesive strips
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-08-15 (Estimated); Primary Completion 2021-12-20 (Estimated); Study Completion 2022-06-20 (Estimated)

PRIMARY OUTCOMES:
Vancouver Scar Scale | 3 months after surgical wound healing
  Vancouver scar scale includes four items toward evaluation of observable aspects of the scar. Each item is rated with 4-6 possible points.

SECONDARY OUTCOMES:
Patient Scar Assessment Scale | From surgical wound healed to 6 months later
  In scar dressing group, patient scar assessment scale consists of 6 questions. Each question is rated from 1 to 10. 1 is the best and 10 reflects the worst.
Incidence of incision site complication | From surgical wound healed to 6 months later
  Percentage of the population suffering from surgical scar-related complications are analyzed, especially the ones toward scar dressing.
Patient satisfaction | 3 months after surgical wound healing
  In scar dressing group, patients are asked with serial questions to rate satisfaction toward scar dressing on a numeric rating scale. 1 means the most unsatisfaction and 10 means the most satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hsieh Chang, Prof., Study Chair — Chang Gung Medical Foundation

IPD SHARING:
Plan to Share IPD: No